CLINICAL TRIAL: NCT01966497
Title: Observational Study of Patients Older Than 60 Years and With Acute Myeloblastic Leukemia Who Are Administered Standard Chemotherapy Based on Idarubicine-cytarabine
Brief Title: Observational Study of Patients Older Than 60 Years With Acute Myeloblastic Leukemia
Acronym: ALFA1200
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI11020
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Acute Myeloblastic Leukemia; Aged Higher Than 60 Years Old
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Core study therapy: * idarubicin for both induction and consolidation courses
  * if Cr, two cycles of IDAC alone (1.5g/m2 per infusion every 12hours, on D1, 3 and 5 of each cycle)

SUMMARY:
The main objective of this observational survey is to estimate the incidence, the typology, and the evolution of patients with acute myelobalstic leukemia, aged more than 60 years old. In this age group (aged more than 60y), three groups of patients with very different response rates and late outcome can be delineated with specific standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or more
* With a morphologically proven diagnosis of AML according to WHO 2008 classification
* Not previously treated for AML
* Signed informed consent.

Exclusion Criteria:

* APL in the WHO classification.
* Ph1-positive AML or prior Ph1-positive disease
* AML evolving from a prior MPN in the WHO 2008 classification.
* Prior tumor, if not stable for at least two years, except in-situ carcinoma and skin carcinoma
* ECOG Performance Status Score > 3
* Positive serology for HIV or HTLV1, or active viralinfection for HBV and HBC.
* Severe uncontrolled infection at inclusion time.
* Psychiatric disease or an history of non-complianceto medical regimens or patients considered potentially unreliable.
* Absence of Health Care Insurance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital admissions from the participating centres
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-11 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of failures | 9 months
  failures include
  * resistant disease defined according to the IWG AML response criteria
  * hypoplastic marrow after D42 and absence of myeloidrecovery
  * early relapse up to 9 months from CR : Either AML relapse as in the IWG classification or MDS relapse

SECONDARY OUTCOMES:
response rate | 9 months
relapse rate | within 2 years after inclusion
  Either AML relapse as in the IWG classification
  - Or MDS relapse defined for this study as follows: (i) Persistent cytopenias, if unexplained by other cause, and (ii) myelodysplastic marrow with less than 20% marrow blasts in two samples taken 3 months apart
overall survival | within 2 years after inclusion
adverse events | within 2 years after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Avicenne, Bobigny, Île-de-France Region, France

REFERENCES:
- [Derived] Gardin C, Pautas C, Fournier E, Itzykson R, Lemasle E, Bourhis JH, Ades L, Marolleau JP, Malfuson JV, Gastaud L, Raffoux E, Lambert J, Braun T, Thomas X, Chantepie S, Cluzeau T, de Botton S, Berthon C, Boissel N, Duployez N, Terre C, Peffault de Latour R, Michallet M, Celli-Lebras K, Preudhomme C, Dombret H. Added prognostic value of secondary AML-like gene mutations in ELN intermediate-risk older AML: ALFA-1200 study results. Blood Adv. 2020 May 12;4(9):1942-1949. doi: 10.1182/bloodadvances.2019001349. PMID 32380535